CLINICAL TRIAL: NCT04703478
Title: RespiraConNosotros: Creation and Implementation of a Mobile Application for the Rehabilitation of Patients With Respiratory Sequelae of the SARS-CoV-2 (COVID-19)
Brief Title: RespiraConNosotros:a Mobile Application for COVID-19 Respiratory Rehabilitation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Beatriz-María Bermejo-Gil, Professor, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CovidSal02
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: respiration disorders; telerehabilitation; breathing exercises; complications
MeSH Terms: conditions — COVID-19; Respiration Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Implementation of a mobile application for the rehabilitation of patients with respiratory sequelae of COVID-19
  Interventions: Other: Breathing exercise

INTERVENTIONS:
Other: Breathing exercise — Participants will carry out a breathing exercise program through the RespiraConNosotros mobile application. They will be asked to carry out the proposed exercises with a frequency of 3 times a week for 3 months.

SUMMARY:
Platform with a mobile application to encourage the performance of respiratory exercises, controlled and supervised by physiotherapists. It also includes recommendations, frequently asked questions and the possibility of contacting by chat or video calls with experts to solve possible doubts.

Currently, the application is ready for use, the registration of users and professionals is enabled and have 20 exercises divided into three intensity levels.

It is available for all platforms (PC, ANDROID, iOS). presents a simple deployment, accessible to the entire population and does not require installation.

In the future, investigators will include more languages, a greater variety of exercises and even other types of therapies. Investigators will also carry out the adaptation to functional diversity with subtitles and voice commands.

ELIGIBILITY:
Inclusion Criteria:

* Respiratory affectation diagnosis
* Internet access to run the application

Exclusion Criteria:

* Presence of contraindications to physical exercise or the lack of comprehensive ability to access the application will be considered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-20 (Estimated); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
Rating of perceived exertion (Borg Scale) | 10 minutes.
  Scale from 1-10 points. Where number 1 means very light activity and 10, represents an extreme intensity of activity.
Level of satisfaction and acceptability. | 20 minutes.
  A Likert-type scale will be used. 1-Not Satisfied to 5-Extremely satisfied.
St. George's Respiratory Questionnaire, SGRQ | 40 minutes.
  scale from 0-100 points.Where higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Age | 2 minutes.
  The date of birth will be registered in order to calculate the age of the participant.
Sex | 2 minutes.
  Participant's sex will be registered
Diagnosis of respiratory pathology | 2 minutes.
  Participant's diagnosis will be registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Ines Llamas-Ramos, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided